CLINICAL TRIAL: NCT04072835
Title: The NODE-303 Study: Multi-Centre, Multi-National,Open Label, Safety Study of Etripamil Nasal Spray for Patients With Paroxysmal Supraventricular Tachycardia.
Brief Title: Safety Study of Etripamil Nasal Spray for Patients With Paroxysmal Supraventricular Tachycardia. NODE-303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NODE-303
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Paroxysmal Supraventricular Tachycardia
Keywords: PSVT
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etripamil NS (Experimental): Participants self-administered etripamil NS 70 mg. After implementation of protocol amendment 2.1 (16 March 2021), participants had the option to administer a second dose of etripamil 70 mg 10 minutes after the first dose, if PSVT symptoms persisted
  Interventions: Drug: Etripamil NS
- Not Treated (No Intervention): Participants not treated with etripamil NS for a PSVT episode.

INTERVENTIONS:
Drug: Etripamil NS — Participants were provided with an ambulatory Cardiac Monitoring System (CMS) to help document PSVT episodes. The CMS was self-applied by the participant, when PSVT symptoms begin. Participants self-administered etripamil NS if vagal maneuver was ineffective. After implementation of protocol amendment 2.1, participants had the option to administer a second dose of etripamil 70 mg 10 minutes after the first dose, if symptoms persisted. After an episode of PSVT where drug was administered, the participant returned to the investigative site for a study visit and was given the option to continue in NODE-303 and manage up to three subsequent episodes of PSVT with etripamil NS for a maximum of four episodes.
  Other Names: MSP-2017
  Arms: Etripamil NS

SUMMARY:
NODE-303 was a multi-center, open label study to evaluate the safety of etripamil NS in participants with Paroxysmal Supraventricular Tachycardia (PSVT). Participants were provided with an ambulatory Cardiac Monitoring System (CMS) to help document PSVT episodes. The CMS was self-applied by the participant, when they felt the onset of PSVT symptoms. Participants self-administered etripamil NS if vagal maneuver was ineffective. After an episode of PSVT where study drug was administered, the participant returned to the investigative site and had the option to continue in NODE-303 and manage up to three subsequent episodes of PSVT with etripamil NS for a maximum of four episodes.

DETAILED DESCRIPTION:
NODE-303 was a multi-center, open label study to evaluate the safety of etripamil NS in participants with PSVT. Participants were provided with an ambulatory CMS to help document PSVT episodes. The CMS was self-applied by the participant, when they felt the onset of PSVT symptoms. Participants self-administered etripamil NS 70 mg if vagal maneuver (VM) was ineffective. Approximately 2 years after study initiation, a protocol amendment was implemented to allow participants to administer a second dose of etripamil 70 mg 10 minutes after the first dose, if PSVT symptoms persisted. After an episode of PSVT where study drug was administered, the participant returned to the investigative site and had the option to continue in NODE-303 and manage up to three subsequent episodes of PSVT with etripamil NS for a maximum of four episodes.

The study included:

A Screening Visit during which the Investigator verified that the participant met the eligibility criteria of the NODE-303 study, obtained the signed informed consent, took blood and urine for laboratory evaluations, and conducted other screening procedures. The informed consent for NODE-303 was applicable for the initial and all subsequent PSVT episodes. A Baseline Visit during which the site confirmed eligibility, concomitant medications, trained the participant on study procedures, and gave the participant study drug, participant reported outcome (PRO) materials, and the CMS materials. A Treatment Period during which the participant completed the monthly PRO survey, self-identified symptoms of PSVT, used the CMS during 60 minutes, performed a VM, and self-administered etripamil NS if the symptoms did not resolve after the VM. Participants could be contacted during this period for reminders and training on what to do during a PSVT episode. Participants also completed a per episode survey after any PSVT episode they experience. During the Treatment Period, Follow-up Visits occurred at the study site up to 14 days after each episode of PSVT treated with etripamil NS, and during which the Investigator evaluated the results of the last usage of etripamil NS and reassessed participant's eligibility to continue in the study based on study inclusion and exclusion criteria. Participants who were eligible to continue in the study received additional study medication.

A Final Study Visit occurred when a participant discontinued or withdrew from the study, or when the overall study was completed, or the participant had completed the maximum number of doses. NODE-303 continued until enough documented self-administrations of etripamil NS were included in the safety database to meet regulatory requirements for the etripamil NS development program. The common study end date (CSED) for the entire study depended on the rate of accrual of the primary endpoint, unique participants with an episode. When the criteria for concluding the study were met, the Sponsor announced the CSED for the entire study and sites were informed in advance to schedule all final participant visits prior to the CSED.

ELIGIBILITY:
Inclusion Criteria:

A participant was eligible for study participation if they met all of the following criteria:

1. Had been diagnosed with PSVT by a medical professional, and reported having at least one previous episode of PSVT. For clarity, PSVT referred to episodic Supraventricular Tachycardia (SVT) that included the atrioventricular (AV) node as a critical part of reentrant circuit.
2. Was at least 18 years of age;
3. Signed NODE-303 written informed consent
4. Women of childbearing potential had to be willing to use at least 1 form of contraception during the trial, and had to be willing to discontinue from the study should they have become or planned to become pregnant. Postmenopausal females were defined as having amenorrhea for at least 12 months prior to Screening without an alternative medical cause.
5. Willing and able to comply with study procedures

Exclusion Criteria:

A participant was excluded from the study if they met any of the following criteria:

1. Participants with only a history of atrial arrhythmia that did not involve the atrioventricular (AV) node as part of the tachycardia circuit (e.g. atrial fibrillation, atrial flutter, intra-atrial tachycardia) were not eligible. Participants with a history of these tachycardias who were also diagnosed with PSVT were eligible.
2. History of allergic reaction to verapamil
3. Current therapy with digoxin, or any Class I or III antiarrhythmic drug. Participants could be eligible if these drugs were stopped at least five half-lives before the administration of etripamil NS. The only exception was amiodarone which had to be stopped 30 days before enrollment.
4. History or evidence of ventricular pre-excitation, e.g., delta waves, Wolff- Parkinson-White syndrome
5. History or evidence of a second- or third-degree AV block
6. History or evidence of severe ventricular arrhythmia (e.g., torsades de pointes, ventricular fibrillation, or sustained ventricular tachycardia).
7. Symptoms of congestive heart failure New York Heart Association Class II to IV
8. SBP < 90 mmHg at Screening, Baseline or any Follow-up Visit.
9. Severe symptoms of hypotension experienced during PSVT episodes.
10. Significant physical or psychiatric condition including alcoholism or drug abuse, which, in the opinion of the Investigator, could jeopardize the safety of the participant, or impede the participant's capacity to follow the study procedures
11. History of syncope due to an arrhythmic etiology at any time, or history in last 5 years of unexplained syncope
12. Was pregnant or breastfeeding
13. Previously enrolled in a clinical trial for etripamil and received study drug or participation in any clinical trial for other investigational products or medical devices within 30 days of Screening.
14. History of Acute Coronary Syndrome (ACS) or stroke within 6 months of screening
15. Evidence of renal dysfunction as determined by an estimated glomerular filtration rate assessed at the Screening Visit as follows:

    1. <60mL/min/1.73m2 for participants <60 years of age;
    2. <40mL/min/1.73m2 for participants ≥60 and <70 years of age
    3. <35mL/min/1.73m2 for participants ≥70 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Plat, MD, Study Director — Milestone Pharmaceuticals
Locations (124):
- United States (61):
  - 1077, Gilbert, Arizona
  - 1121, Fremont, California
  - 1035, Stanford, California
  - 1023, Vista, California
  - 1083, West Hills, California
  - 101, Littleton, Colorado
  - 1010, Bridgeport, Connecticut
  - 1066, Trumbull, Connecticut
  - 1042, Bradenton, Florida
  - 1106, Daytona Beach, Florida
  - 1107, Edgewater, Florida
  - 1032, Hialeah, Florida
  - 1026, Miami, Florida
  - 1055, Miami, Florida
  - 1064, Naples, Florida
  - 1071, North Miami Beach, Florida
  - 1009, Orlando, Florida
  - 1060, Saint Augustine, Florida
  - 1022, Cumming, Georgia
  - 137, Macon, Georgia
  - 1115, Coeur d'Alene, Idaho
  - 1045, Peoria, Illinois
  - 149, Fort Wayne, Indiana
  - 1025, West Des Moines, Iowa
  - 1008, Monroe, Louisiana
  - 1007, Salisbury, Maryland
  - 1078, Boston, Massachusetts
  - 166, Lansing, Michigan
  - 119, Rochester, Minnesota
  - 1093, Saint Paul, Minnesota
  - 1099, Kansas City, Missouri
  - 1134, Elmer, New Jersey
  - 1133, Haddon Heights, New Jersey
  - 114, New York, New York
  - 1021, Southampton, New York
  - 129, Charlotte, North Carolina
  - 1065, Charlotte, North Carolina
  - 1079, Mount Airy, North Carolina
  - 1018, Statesville, North Carolina
  - 1024, Canton, Ohio
  - 123, Cincinnati, Ohio
  - 142, Columbus, Ohio
  - 1086, Oklahoma City, Oklahoma
  - 1123, Corvallis, Oregon
  - 1031, Hershey, Pennsylvania
  - 1082, Wyomissing, Pennsylvania
  - 105, Yardley, Pennsylvania
  - 1097, York, Pennsylvania
  - 122, Rapid City, South Dakota
  - 1062, Jackson, Tennessee
  - 1012, Memphis, Tennessee
  - 1047, Austin, Texas
  - 1092, Austin, Texas
  - 1016, Fort Worth, Texas
  - 1017, Houston, Texas
  - 1048, Plano, Texas
  - 1014, San Antonio, Texas
  - 1004, Riverton, Utah
  - 117, Lynchburg, Virginia
  - 1076, Richmond, Virginia
  - 0116, Richmond, Virginia
- Argentina (18):
  - 5106, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - 5117, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - 5112, Mar del Plata, Buenos Aires
  - 5105, Mar del Plata, Buenos Aires
  - 5115, Quilmes, Buenos Aires
  - 5122, Ramos Mejía, Buenos Aires
  - 5110, San Nicolás de los Arroyos, Buenos Aires
  - 5129, Buenos Aires
  - 5125, Buenos Aires
  - 5134, Corrientes
  - 5116, Córdoba
  - 5123, Córdoba
  - 5118, Córdoba
  - 5102, La Plata
  - 5132, Rosario
  - 5109, Salta
  - 5130, San Nicolás
  - 5124, Temperley
- Brazil (21):
  - 5221, Belo Horizonte, REG1
  - 5217, Brasília, REG1
  - 5215, Campinas, REG1
  - 5222, Canoas, REG1
  - 5207, Curitiba, REG1
  - 5227, Juiz de Fora, REG1
  - 5209, Recife, REG1
  - 5214, Salvador, REG1
  - 5219, Santo André, REG1
  - 5212, São José do Rio Preto, REG1
  - 5220, São Paulo, REG1
  - 5225, São Paulo, REG1
  - 5205, Uberlândia, REG1
  - 5228, Belo Horizonte
  - 5202, Campinas
  - 5201, Goiânia
  - 5229, Jaú
  - 5235, Rio de Janeiro
  - 5232, São Paulo
  - 5204, Tatuí
  - 5231, Votuporanga
- Canada (18):
  - 2017, Kelowna, British Columbia
  - 2010, North Vancouver, British Columbia
  - 2019, Saskatoon, British Columbia
  - 2018, Surrey, British Columbia
  - 212, Vancouver, British Columbia
  - 213, Victoria, British Columbia
  - 215, Cambridge, Ontario
  - 202, Hamilton, Ontario
  - 2006, Oshawa, Ontario
  - 2001, Ottawa, Ontario
  - 2011, Greenfield Park, Quebec
  - 2020, Lévis, Quebec
  - 205, Montreal, Quebec
  - 203, Montreal, Quebec
  - 2014, Québec, Quebec
  - 2002, Saint-Jean-sur-Richelieu, Quebec
  - 2003, Saint-Jérôme, Quebec
  - 201, Sherbrooke, Quebec
- Colombia (6):
  - 5409, Armenia
  - 5404, Barranquilla
  - 5408, Bucaramanga
  - 5401, Medellín
  - 5407, Punta de Cartagena
  - 5403, San Gil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorian P, Alings M, Coutu B, Ip JE, Martinez FA, Piccini JP, Stambler BS, Sheikh M, Shardonofsky S, Bharucha DB, Camm AJ. Self-Administered Etripamil Nasal Spray Slows Ventricular Rate in Patients With Atrial Fibrillation: A Post Hoc Analysis of the NODE-303 Study. J Cardiovasc Electrophysiol. 2026 Feb 10. doi: 10.1111/jce.70287. Online ahead of print. PMID 41668514
- [Derived] Ip JE, Coutu B, Ip JH, Noseworthy PA, Parody ML, Rafii F, Sears SF, Singh N, Stambler BS, Tahirkheli NK, Agudelo-Uribe J, Hu D, Shardonofsky S, Sheikh MB, Holz A, Bharucha DB, Camm AJ. Etripamil Nasal Spray for Recurrent Paroxysmal Supraventricular Tachycardia Conversion: Results From the NODE-303 Open-Label Study. J Cardiovasc Electrophysiol. 2025 Nov;36(11):2990-3003. doi: 10.1111/jce.70086. Epub 2025 Sep 11. PMID 40931676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To enroll participants in the study, a diagnosis of PSVT by a medical professional and history of at least one previous episode of PSVT were required. The first participant was enrolled on September 23, 2019 and the last participant was enrolled on October 27, 2022.
Pre-assignment Details: Participants had to meet all inclusion criteria and none of the exclusion criteria to be enrolled in the study. At baseline, the participants received the CMS, the study drug, and instructions on what to do when they started to feel the symptoms of PSVT.
Groups:
- All Participants: Participants self-administered etripamil NS 70 mg and after the implementation of protocol amendment 2.1, the participants had the option to administer a second dose of etripamil 70 mg 10 minutes later, if PSVT symptoms persisted.
  Considering this is an event-driven study, not all participants experienced a PSVT and could administered the study drug before the study was completed. This arm includes all participants that were enrolled in the study.
Period: Overall Study
Arm/Group | All Participants
Started (Enrolled in the study but not all have experienced a PSVT episode and administered the study drug before the end of the study.) | 1116
Participants Who Completed the Study With at Least 1 Treated Perceived PSVT Episode | 503
Participants Who Treated 1 Perceived PSVT Episode in the Study | 220
Participants Who Treated 2 Perceived PSVT Episodes in the Study | 118
Participants Who Treated 3 Perceived PSVT Episodes in the Study | 62
Participants Who Treated 4 Perceived PSVT Episodes in the Study | 103
Completed | 103
Not Completed | 1013
Not completed — Overall trial ended | 603
Not completed — Ablation | 97
Not completed — Withdrawal of consent | 66
Not completed — Physician Decision | 50
Not completed — Lost to Follow-up | 39
Not completed — Participant no longer meets the inclusion/exclusion criteria | 38
Not completed — Participant wanted to try other therapy or treatment | 34
Not completed — Adverse Event | 25
Not completed — Participant non-compliance / Protocol violation(s) | 25
Not completed — Death | 11
Not completed — Participant felt the drug did not work | 8
Not completed — Participant tolerability | 5
Not completed — Missing | 5
Not completed — Participant withdrawn due to COVID-19 situation | 4
Not completed — Pregnancy | 3

BASELINE CHARACTERISTICS:
Population: Overall population
Groups:
- All Participants: Participants self-administered etripamil NS 70 mg and after the implementation of protocol amendment 2.1, the participants had the option to administer a second dose of etripamil 70 mg 10 minutes later, if PSVT symptoms persisted.
  Considering this is an event-driven study, not all participants experienced a PSVT and could administered the study drug before the study was completed. This arm/group includes all participants that were enrolled in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 1116
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at informed consent signed | 54.3 (14.0)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Not all participants reported the age at first diagnostic of PSVT
  years
    Age at first diagnosis of PSVT: number analyzed (Participants) | 875
    Age at first diagnosis of PSVT | 48.3 (16.2)
Age, Customized [Count of Participants; unit: Participants]
  Age at informed consent signed: 18 to < 60 years | 695
  Age at informed consent signed: 60 to < 70 years | 263
  Age at informed consent signed: ≥ 70 years | 158
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 762
  Male | 354
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 396
  Not Hispanic or Latino | 696
  Unknown or Not Reported | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 57
  White | 913
  More than one race | 0
  Unknown or Not Reported | 106
Weight [Mean (Standard Deviation); unit: Kg] | 82.3 (21.5)
Height [Mean (Standard Deviation); unit: cm] — Population: Not all participants reported the height
  cm
    number analyzed (Participants) | 1111
    (all) | 167.2 (9.4)
Time since first PSVT diagnosis [Mean (Standard Deviation); unit: years] — Population: Not all participants reported the time since first PSVT diagnosis
  years
    number analyzed (Participants) | 875
    (all) | 6.2 (8.9)
Number of participant-reported PSVT episodes in the past year [Mean (Standard Deviation); unit: episodes] — Population: Not all participants reported PSVT episodes in the past year
  episodes
    number analyzed (Participants) | 1064
    (all) | 8.6 (16.5)
Number of participant-reported emergency department visits since diagnosis [Mean (Standard Deviation); unit: emergency department visits] — Population: Not all participants reported emergency department visit
  emergency department visits
    number analyzed (Participants) | 647
    (all) | 3.5 (6.3)
Number of participant-reported urgent care visits since diagnosis [Mean (Standard Deviation); unit: urgent care visits] — Population: Not all participants reported urgent care visits
  urgent care visits
    number analyzed (Participants) | 168
    (all) | 5.0 (11.2)
Number of participant-reported visits to doctor's office since diagnosis [Mean (Standard Deviation); unit: visits to doctor's office] — Population: Not all participants reported visits to doctor's office
  visits to doctor's office
    number analyzed (Participants) | 324
    (all) | 5.0 (10.2)
Number of participant-reported visits to the arrhythmia clinic / day hospital since diagnosis [Mean (Standard Deviation); unit: visits to the arrhythmia clinic/day hosp] — Population: Not all participants reported visits to the arrhythmia clinic/day hospital
  visits to the arrhythmia clinic/day hosp
    number analyzed (Participants) | 61
    (all) | 5.0 (13.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events for Self-administered Etripamil NS Outside of the Clinical Setting.
Description: Number of participants with any adverse events experienced from baseline up to the final study visit including the treatment of up to 4 perceived PSVT episodes.
Time Frame: From Baseline until a maximum of 4 episodes of perceived PSVT are treated with study drug, up to a maximum duration of 40 months.
Population: The Safety Population includes all participants who self-administered any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Etripamil: Participants self-administered etripamil NS 70 mg and after the implementation of protocol amendment 2.1, the participants had the option to administer a second dose of etripamil 70 mg 10 minutes later, if PSVT symptoms persisted.
  Only participants that received etripamil are included in this group. All adverse events reactions were included regardless of treatment-emergent status and causality assessment
Arm/Group | Etripamil
Number analyzed (Participants) | 503
Participants | 324

2. Secondary Outcome: Time to Conversion
Description: Kaplan-Meier estimates of time to conversion up to 60 minutes after etripamil administration for adjudicated conversion of confirmed episodes of PSVT to SR (Sinus Rhythm) reported at Follow-up Visit 1.
Time Frame: Time to conversion up to 60 minutes after etripamil administration.
Population: The Efficacy Population includes participants who received study drug for an event confirmed as PSVT by the Sponsor's medical review of the ECG CMS data.
Measure: Median (95% Confidence Interval); unit: minutes
Groups:
- Etripamil: Participants self-administered etripamil NS 70 mg and after the implementation of protocol amendment 2.1, the participants had the option to administer a second dose of etripamil 70 mg 10 minutes later, if PSVT symptoms persisted.
  Only participants that received etripamil for a confirmed PSVT episode are included in this group.
Arm/Group | Etripamil
Number analyzed (Participants) | 231
minutes | 17.7 [13.9 to 26.2]

ADVERSE EVENTS:
Time Frame: From Baseline until a maximum of 4 episodes of perceived PSVT are treated with study drug, up to a maximum duration of 40 months.
Description: Adverse Events (including All-Cause Mortality, Serious Adverse Events and Other (not including Serious) Adverse Events are reported for participants in the safety population (i.e., enrolled participants who took at least 1 dose of study drug and are the "population at risk"; N=503). For completeness, participants who were enrolled in the study but did not treat a PSVT episode with study drug are included under the Not Treated column
Groups:
- Etripamil: Participants self-administered etripamil NS 70 mg and after the implementation of protocol amendment 2.1, the participants had the option to administer a second dose of etripamil 70 mg 10 minutes later, if PSVT symptoms persisted.
- Not Treated: Participants not treated with etripamil NS. Participants were still waiting for their first perceived PSVT episode when this event-driven study was ended by the sponsor.
Arm/Group | Etripamil | Not Treated
All-Cause Mortality (participants affected / at risk) | 4/503 | 7/613
Serious Adverse Events (participants affected / at risk) | 34/503 | 22/613
Other Adverse Events (participants affected / at risk) | 237/503 | 32/613
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etripamil (N=503) | Not Treated (N=613)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Corona virus infection (Infections and infestations) | 2 | 5
Osteomyelitis (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Septic shock (Infections and infestations) | 1 | 0
Device related Thrombosis (General disorders) | 1 | 0
Viral vasculitis (Infections and infestations) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Gastric fistula (Gastrointestinal disorders) | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etripamil (N=503) | Not Treated (N=613)
Headache (Nervous system disorders) | 28 (40) | 4 (5)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 153 (235) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 72 (96) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 68 (98) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 41 (49) | 0 (0)
Corona virus infection (Infections and infestations) | 28 (30) | 26 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT04072835/Prot_002.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT04072835/SAP_001.pdf